CLINICAL TRIAL: NCT01457261
Title: A Study of the Pharmacokinetics and Deposition of Inhaled Salbutamol in Patients With Idiopathic Pulmonary Fibrosis (TOPICAL-IPF)
Brief Title: IPF Drug Deposition Study
Acronym: TOPICAL-IPF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHIPF02; 2011-000336-29 (EudraCT Number)
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: interstitial lung disease; drug deposition; lung imaging; respiratory
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Partical size 1 (Experimental): Monodisperse particle delivered with radiolabel
  Interventions: Drug: Salbutamol
- Particle size 2 (Experimental): Monodisperse particle delivered with radiolabel
  Interventions: Drug: Salbutamol
- Nebulised salbutamol (Experimental): Polydisperse particle via a nebuliser
  Interventions: Drug: Salbutamol
- Salbutamol MDI (Experimental): Unlabelled salbutamol via a metered dose inhaler
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Salbutamol — Radiolabelled salbutamol to be administered as a monodisperse particle via a spinning top aerosol generator or else as a polydisperse mist via a nebuliser or metered dose inhaler.
  Other Names: Ventolin

SUMMARY:
Idiopathic pulmonary fibrosis is a relentlessly progressive disease that is responsible for the deaths of over 5000 people in the UK each year. At present, despite a dramatic increase in clinical trials in the last decade, there are no licensed treatments for IPF. The pathogenesis of the condition remains incompletely understood, nonetheless there is good evidence to suggests that the condition arises as the consequence of an aberrant wound healing response in genetically susceptible individuals. Basic science research into IPF has identified a wide range of potential treatment targets. However, in many cases developing compounds to act against these targets, because of their role in normal wound healing, is limited by the possibility of major systemic side effects.

The lung is highly amenable to topical therapy in the form of inhaled drug preparations and this route is utilised in the treatment of the majority of respiratory disease. The inhaled route offers a number of important potential advantages for administration of therapy to patients with IPF. Firstly, by limiting systemic exposure to drugs, the inhaled route offers the potential for achieving higher lung doses of drugs that might otherwise cause systemic toxicity. Secondly, inhaled treatment may more effectively reach the areas of abnormality in IPF, namely the hyperplastic epithelium and the underlying fibroblastic foci. Thirdly, the inhaled route offers an alternative to parenteral administration of compounds that are poorly absorbed through the gastro-intestinal tract e.g. monoclonal antibodies. It should be noted however, that the fibrosis in IPF develops peripherally involving the alveolar interstitium and the terminal bronchioles. Furthermore, the disease causes architectural destruction and distortion of the lung that is liable to alter the normal laminar flow of air (and inhaled particles) through the bronchial tree. It is therefore, by no means certain that it is possible to deliver inhaled therapies directly to regions of fibrosis in IPF.

The feasibility of delivering inhaled drugs in IPF has not been previously studied. This research by assessing the effect of particle size on inhaled particle deposition and by relating to this the pharmacokinetic profile of salbutamol aims to validate the potential of the inhaled route in IPF. This study is an important precursor to the development of specific topical therapies for patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of definite or probable idiopathic pulmonary fibrosis as defined by the ATS/ERS consensus criteria

Exclusion Criteria:

* co-existent respiratory disease
* use of B2 agonists in preceding two weeks
* DLco and/or FVC falling outside the criteria for either mild or severe IPF.
* Ongoing involvement in clinical trials assessing novel IPF therapies.
* Previous adverse reaction to short or long acting β2 agonist.
* Pregnancy or active breast feeding
* Any contraindication to taking inhaled beta-2 adrenoceptor agonists (especially salbutamol) as listed in the British National Formulary will not be entered into this study.
* an acute respiratory exacerbation requiring emergency room treatment and/ or hospitalisation within four weeks of visit 1 (screening visit)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Total lung deposition | 5 minutes post administation
  Effect of particle size and delivery device will be assessed by measuring total lung deposition of radio-labelled particles on scintegraphic images

SECONDARY OUTCOMES:
Serum salbutamol change | 0 - 6 hours
  Pharmacokinetics of inhaled drug absorbtion
Urinary salbutamol concentration | 0-8 hours
  Measurement of pharmacokinetics of salbutamol absorbtion through measurement of urinary excretion
Penetration index | 5 minutes post administration
  Measure of pattern of drug distribution (procximal versus distal lung) as determined by lung scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Toby M Maher, MB PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom

REFERENCES:
- [Background] Maher TM, Wells AU, Laurent GJ. Idiopathic pulmonary fibrosis: multiple causes and multiple mechanisms? Eur Respir J. 2007 Nov;30(5):835-9. doi: 10.1183/09031936.00069307. PMID 17978154
- [Background] Usmani OS, Biddiscombe MF, Underwood SR, Barnes PJ. Characterization of the generation of radiolabeled monodisperse albuterol particles using the spinning-top aerosol generator. J Nucl Med. 2004 Jan;45(1):69-73. PMID 14734675
- [Background] Usmani OS, Biddiscombe MF, Barnes PJ. Regional lung deposition and bronchodilator response as a function of beta2-agonist particle size. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1497-504. doi: 10.1164/rccm.200410-1414OC. Epub 2005 Sep 28. PMID 16192448
- [Derived] Usmani OS, Biddiscombe MF, Yang S, Meah S, Oballa E, Simpson JK, Fahy WA, Marshall RP, Lukey PT, Maher TM. The topical study of inhaled drug (salbutamol) delivery in idiopathic pulmonary fibrosis. Respir Res. 2018 Feb 6;19(1):25. doi: 10.1186/s12931-018-0732-0. PMID 29409488